CLINICAL TRIAL: NCT04264975
Title: Utilization of Microbiome as Biomarkers and Therapeutics in Immuno-Oncology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sook Ryun Park, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0608
Record Dates: First submitted 2020-01-02; First posted 2020-02-11 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Solid Carcinoma
Keywords: immuno-oncology; immunotherapy; biomarker; fecal microbiota transplantation (FMT); microbiome
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is an open label, single-center, non-randomized clinical trial on utilization of microbiome as biomarkers and therapeutics in immuno-oncology.
  This research consists of two parts:
  part 1: development of microbiome biomarkers for immuno-oncology part 2: proof-of-concept trial on the fecal microbiota transplantation in patients who are being treated with immunotherapy for advanced solid tumor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal microbiota transplantation (Experimental): Fecal microbiota transplantation in patients who have advanced solid cancer with primary (group 1) or secondary resistance (group 2) to immuno-oncology
  Interventions: Procedure: fecal microbiota transplantation

INTERVENTIONS:
Procedure: fecal microbiota transplantation — Fecal microbiota transplantation (FMT) is the administration of a solution of fecal matter from a donor into the intestinal tract of a recipient in order to directly change the recipient's microbial composition and confer a health benefit
  Other Names: FMT

SUMMARY:
This is an open label, single-center, non-randomized clinical trial on utilization of microbiome as biomarkers and therapeutics in immuno-oncology.

This research consists of two parts:

part 1: development of microbiome biomarkers for immuno-oncology part 2: proof-of-concept trial on the fecal microbiota transplantation in patients who are being treated with immunotherapy for advanced solid tumor

ELIGIBILITY:
Part 1: development of microbiome biomarkers

<Inclusion Criteria:> 1.Patients with pathologically confirmed solid cancer who are being treated with immunotherapy or are going to receive immunotherapy

1. Age ≥ 19 years old
2. Eastern Cooperative Oncology Group performance status 0-2
3. Measurable or evaluable lesion(s) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

<Exclusion Criteria>

1. A history of other cancers requiring treatment within the recent 3 years (excepting treated basal or squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, breast, or stomach)
2. A history of active primary immunodeficiency
3. Active infection including tuberculosis or Human Immunodeficiency Virus (HIV)
4. Autoimmune disease (excepting type 1 diabetes mellitus, hypothyroidism requiring hormone replacement therapy only, skin disease not requiring systemic therapy (such as vitiligo, psoriasis or alopecia)
5. Patients who are receiving immunosuppressive medications (excepting topical steroids, systemic steroid ≤10 mg/day prednisone or equivalents, or a brief course of steroids for prophylaxis (e.g., hypersensitivity reaction)

   --------------------------------------------------------------------------------------------

part 2: proof-of-concept trial on the fecal microbiota transplantation in patients who are being treated with immunotherapy for solid cancers

<Inclusion Criteria for donors>

1. Patients who have partial or complete response to immunotherapy at the time of stool donation
2. No history of exposure to HIV or hepatitis virus within the previous 12 months
3. No history of international travel within previous 6 months to areas of high risk of travelers' diarrhea
4. No current communicable disease
5. No household members with active gastrointestinal infection
6. No history of inflammatory bowel disease
7. No recent intake of potential allergenic foods that are known to cause hypersensitivity in a recipient (such as peanut)

<Inclusion criteria for recipients>

1. Patients without contraindications for colonoscopy such as suspected bowel perforation, acute diverticulitis, or fulminant colitis
2. Patients who have disease progression to immunotherapy as one of the following two patterns:

2-1) Patients who have disease progression due to primary resistance to immunotherapy

2-2) Patients who have disease progression following disease stabilization due to secondary resistance to immunotherapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 5 years
  the proportion of patients who have a partial or complete response to therapy per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 or immune RECIST(iRECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, M.D, Ph D, Principal Investigator — Asan Medical Center, Ulsan University of College of Medicine
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not planned.